CLINICAL TRIAL: NCT07174622
Title: Real-world Clinical Outcomes in Medicare Patients With Hypertension Treated With Symplicity Renal Denervation Plus Standard of Care Versus Standard of Care in Integrated EHR and Claims Data
Brief Title: Longitudinal Real-world Clinical Outcomes Study on Symplicity Renal Denervation
Acronym: SPYRAL CARE
Status: Recruiting | Type: Observational
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Other Study IDs: 14467
Record Dates: First submitted 2025-09-11; First posted 2025-09-16 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-09

CONDITIONS: Hypertension; Cardiovascular Diseases; Vascular Diseases
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Symplicity RDN + SOC: Medicare patients on a stable antihypertension medication regimen and received RDN with a Symplicity RDN system
  Interventions: Device: Renal Denervation (Symplicity Spyral™)
- SOC: Medicare patients on a stable antihypertension medication regimen

INTERVENTIONS:
Device: Renal Denervation (Symplicity Spyral™) — Symplicity Spyral™ multi-electrode renal denervation system
  Groups: Symplicity RDN + SOC

SUMMARY:
This observational study will assess the long-term effectiveness of the RDN procedure for lowering blood pressure in Medicare patients with uncontrolled hypertension. This research will be conducted using de-identified electronic health records (EHR) and administrative health insurance claims data. Patients are enrolled through the submission of claims or encounter data to CMS.

DETAILED DESCRIPTION:
The SPYRAL CARE study is an observational, non-interventional study of the Medicare population with uncontrolled hypertension treated with either the Symplicity RDN system plus standard of care (SOC) or with SOC alone. SOC reflects active management of hypertension. The study will evaluate real-world clinical outcomes by examining deidentified, longitudinal data from administrative health insurance claims linked with EHR. The primary objective is to assess the change in office systolic blood pressure at two years for patients treated with Symplicity RDN plus SOC compared to similar patients receiving SOC alone. The secondary objective is to describe major adverse cardiac events over a two-year period in both groups. The study analysis is subject to a central Institutional Review Board (IRB) review. However, individual hospitals are not engaged in research, and local IRB oversight is not necessary.

ELIGIBILITY:
Inclusion Criteria:

* ≥12 months of history of continuous health plan enrollment with medical and prescription coverage
* Age ≥65 and enrolled in a Medicare plan
* Stable antihypertension regimen and on ≥1 antihypertensive medications
* Diagnosis of uncontrolled hypertension (> 140/90 mm Hg)

Exclusion Criteria:

* A prior RDN procedure
* Diagnosis of secondary hypertension
* Any condition for which RDN is contraindicated

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population will consist of patients enrolled in Medicare and aged 65 and older treated with RDN or on stable antihypertension management in any US location.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Change in Office Systolic Blood Pressure (OSBP) | 2 years
  Change in OSBP at two years relative to baseline between matched treated and comparator cohorts.

SECONDARY OUTCOMES:
Time to Major Cardiovascular Event (MACE) | 2 years
  The secondary outcome is time to MACE over 2 years for the matched treated and comparator cohorts. MACE is defined as the composite of non-fatal stroke, non-fatal myocardial infarction, and all-cause death.

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Secemsky, MD, MSc, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No